CLINICAL TRIAL: NCT03178032
Title: Phase I Trial of DNX-2401 for Diffuse Intrinsic Pontine Glioma Newly Diagnosed in Pediatric Patients.
Brief Title: Oncolytic Adenovirus, DNX-2401, for Naive Diffuse Intrinsic Pontine Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: DNAtrix, Inc. (Industry); Alcyone Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D24-DIPG
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Brainstem Glioma; Neoadjuvant Therapy
Keywords: Diffuse intrinsic pontine gliomas; Oncolytic adenovirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single arm treatment DNX-2401 (Experimental): Single arm receiving virus DNX-2401 infusion after tumor biopsy
  Interventions: Biological: DNX-2401

INTERVENTIONS:
Biological: DNX-2401 — Brain infusion of the virus through the cerebellar peduncle
  Other Names: Delta-24

SUMMARY:
Oncolytic adenovirus for pediatric naive DIPG, to be infused after tumor biopsy through the same trajectory in the cerebellar peduncle.

DETAILED DESCRIPTION:
Diffuse pontine gliomas (DIPG) are one of the most lethal pediatric tumors. All treatment approaches for these tumors have failed, leaving a terrible prospect with median survival under one year, and survival at 5 years virtually of zero. Moreover, most of the long term survivors suffer from long-term side effects of the aggressive treatment. Thus, new therapeutic strategies are required that allow not only for more effective treatments of these tumors but also that defer the severe side effects derived from the current therapeutic choices. DNX-2401 is an oncolytic virus engineered to replicate specifically in tumor cells with an abnormal retinoblastoma (RB) pathway. Moreover, this virus infects cells through integrins, which are more abundant in glioma cells. Here we propose a phase I, unicentric, non-randomized clinical trial to study the safety and potential efficacy of intratumoral administration of DNX-2401 in DIPG. The virus administration will be done after stereotactic tumor biopsy, using the same trajectory, after verification of catheter position with intraoperative MRI. After 3-4 weeks patients will receive standard radiotherapy and/or chemotherapy. The primary objective is to confirm the safety of the target dose known from adults trials. Secondary endpoints are overall survival at 12 months (OS12), percentage of responses and induced immune response against tumor. The follow up includes close monitoring of neurological status, blood tests and brain MRI. If this trial shows evidence of safety and efficacy will propel a multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent OF PATIENT OR PARENTS
2. Patient must be, in the investigator opinion, able to comply with all the protocol procedures.
3. Age 1 - 18 years
4. Negative pregnant blood test in case of fertile women (A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
5. Patient newly diagnosed of DIPG in MRI
6. Lansky Performance Status ≥ 70 before inclusion
7. Lesion considered by the investigator to be accessible for stereotactic biopsy. Lesion location will allow injection without entrance of virus in the ventricular system.
8. No previous treatment for DIPG

Exclusion Criteria:

1. Severe infections or intercurrent medical conditions including, but not limited to, severe renal, hepatic, heart or bone marrow failure, that, on investigator´s criteria, do not allow the inclusion. Patients must be afebrile at baseline [i.e., < 38 degrees (Cº)].
2. Investigational medication in the previous 30 days.
3. Subjects with immunodeficiency, autoimmune conditions or active hepatitis.
4. Any medical or psychological condition that might interfere with the subject's ability to participate if older than 16 years or parents ability when younger than 16, or give informed consent or would compromise the patient's ability to tolerate therapy or any disease that will obscure toxicity or dangerously alter drug metabolism.
5. Tumor with multiple locations or doubt in MRI of a DIPG.
6. Pregnant or breast-feeding females will be excluded, due to the risk for the fetal development of a recombinant virus containing genes related to cellular growth and differentiation.
7. Severe bone marrow hypoplasia.
8. AST (aspartate transaminase) and/or ALT (alanine transaminase)> 3 times over upper normal laboratory level
9. Neutrophils < 1 x 109/L
10. Thrombocytes ≤ 100 x 109/L
11. Hemoglobin < 9g/dl

13. Patients with Li-Fraumeni Syndrome or with a known germ line deficit in the retinoblastoma gene or its related pathways.

14. Vaccinations of any kind within 30 days prior to DNX-2401 administration. 15. Transfusions or medications (G-CSF) to treat pancytopenia or other hematological conditions within 28 days of baseline.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and toxicity of DNX-2401 injected in the cerebellar peduncle | 12 weeks after virus injection
  The trial will look for hematologic and neurologic toxicity (NCI-CTCAE v 4.03).

SECONDARY OUTCOMES:
OS12 | 12 months after virus injection
  Overall Survival at 12 months
Images response | 12 months after virus injection
  Complete/partial response in MRI
QoL | 12 months after virus injection
  measure quality of life baseline assessment and any changes over time
Samples collection | 12 weeks after virus injection
  Collect tumor and blood samples for futures molecular and immune studies.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Gallego, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
During the trail the results will be presented in scientific meetings. After the trial, a paper will be published by the IP

REFERENCES:
- [Result] Alonso MM, Gomez-Manzano C, Bekele BN, Yung WK, Fueyo J. Adenovirus-based strategies overcome temozolomide resistance by silencing the O6-methylguanine-DNA methyltransferase promoter. Cancer Res. 2007 Dec 15;67(24):11499-504. doi: 10.1158/0008-5472.CAN-07-5312. PMID 18089777
- [Result] Jansen MH, Veldhuijzen van Zanten SE, Sanchez Aliaga E, Heymans MW, Warmuth-Metz M, Hargrave D, van der Hoeven EJ, Gidding CE, de Bont ES, Eshghi OS, Reddingius R, Peeters CM, Schouten-van Meeteren AY, Gooskens RH, Granzen B, Paardekooper GM, Janssens GO, Noske DP, Barkhof F, Kramm CM, Vandertop WP, Kaspers GJ, van Vuurden DG. Survival prediction model of children with diffuse intrinsic pontine glioma based on clinical and radiological criteria. Neuro Oncol. 2015 Jan;17(1):160-6. doi: 10.1093/neuonc/nou104. Epub 2014 Jun 5. PMID 24903904
- [Result] Jiang H, Gomez-Manzano C, Aoki H, Alonso MM, Kondo S, McCormick F, Xu J, Kondo Y, Bekele BN, Colman H, Lang FF, Fueyo J. Examination of the therapeutic potential of Delta-24-RGD in brain tumor stem cells: role of autophagic cell death. J Natl Cancer Inst. 2007 Sep 19;99(18):1410-4. doi: 10.1093/jnci/djm102. Epub 2007 Sep 11. PMID 17848677
- [Derived] Gallego Perez-Larraya J, Garcia-Moure M, Labiano S, Patino-Garcia A, Dobbs J, Gonzalez-Huarriz M, Zalacain M, Marrodan L, Martinez-Velez N, Puigdelloses M, Laspidea V, Astigarraga I, Lopez-Ibor B, Cruz O, Oscoz Lizarbe M, Hervas-Stubbs S, Alkorta-Aranburu G, Tamayo I, Tavira B, Hernandez-Alcoceba R, Jones C, Dharmadhikari G, Ruiz-Moreno C, Stunnenberg H, Hulleman E, van der Lugt J, Idoate MA, Diez-Valle R, Esparragosa Vazquez I, Villalba M, de Andrea C, Nunez-Cordoba JM, Ewald B, Robbins J, Fueyo J, Gomez-Manzano C, Lang FF, Tejada S, Alonso MM. Oncolytic DNX-2401 Virus for Pediatric Diffuse Intrinsic Pontine Glioma. N Engl J Med. 2022 Jun 30;386(26):2471-2481. doi: 10.1056/NEJMoa2202028. PMID 35767439
- [Derived] Martinez-Velez N, Garcia-Moure M, Marigil M, Gonzalez-Huarriz M, Puigdelloses M, Gallego Perez-Larraya J, Zalacain M, Marrodan L, Varela-Guruceaga M, Laspidea V, Aristu JJ, Ramos LI, Tejada-Solis S, Diez-Valle R, Jones C, Mackay A, Martinez-Climent JA, Garcia-Barchino MJ, Raabe E, Monje M, Becher OJ, Junier MP, El-Habr EA, Chneiweiss H, Aldave G, Jiang H, Fueyo J, Patino-Garcia A, Gomez-Manzano C, Alonso MM. The oncolytic virus Delta-24-RGD elicits an antitumor effect in pediatric glioma and DIPG mouse models. Nat Commun. 2019 May 28;10(1):2235. doi: 10.1038/s41467-019-10043-0. PMID 31138805